CLINICAL TRIAL: NCT00004866
Title: A Phase II Study of Intravenous DX-8951f Administered Daily for Five Days Every Three Weeks to Patients With Advanced or Recurrent Squamous Cell Cancer of the Cervix
Brief Title: DX-8951f in Treating Women Who Have Advanced or Recurrent Cancer of the Cervix
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067525; DAIICHI-8951A-PRT015; MDA-DM-99247
Record Dates: First submitted 2000-03-07; First posted 2003-01-27 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Cervical Cancer
Keywords: stage III cervical cancer; stage IV cervical cancer; recurrent cervical cancer; cervical squamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — exatecan

INTERVENTIONS:
Drug: exatecan mesylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of DX-8951f in treating women who have advanced or recurrent cancer of the cervix.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of DX-8951f in women with advanced or recurrent squamous cell carcinoma of the cervix.
* Evaluate the quantitative and qualitative toxic effects of this regimen in these patients.
* Evaluate the pharmacokinetics of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive DX-8951f IV over 30 minutes daily for 5 days. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months until death.

PROJECTED ACCRUAL: Approximately 37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced or recurrent squamous cell carcinoma of the cervix not curable by surgery or radiotherapy
* Measurable disease
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT or SGPT no greater than 2 times upper limit of normal (ULN) (5 times ULN if liver metastases present)

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No active congestive heart failure
* No uncontrolled angina
* No myocardial infarction within the past 6 months

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No concurrent serious infection
* No other malignancy within the past 5 years except nonmelanomatous skin cancer
* No other life threatening illness
* No psychosis, mental disability, or incompetence

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent biologic therapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy
* No more than 1 prior chemotherapy regimen (except chemotherapy for radiosensitization)
* No prior camptothecin
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* At least 4 weeks since prior surgery
* No concurrent surgery

Other:

* At least 4 weeks since other prior investigational drugs (including analgesics or antiemetics)
* No other concurrent investigational drugs during or within 28 days after final dose of study drug
* No concurrent drugs that induce or inhibit CYP3A enzyme

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-01; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. DeJager, MD, FACP, Study Chair — Daiichi Sankyo
Locations (6):
- United States (6):
  - St. Luke's-Roosevelt Hospital, New York, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - Ruppert Health Center, Toledo, Ohio
  - Brookview Research, Inc., Nashville, Tennessee
  - Texas Oncology PA (TOPA) at Baylor-Sammons, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas